CLINICAL TRIAL: NCT05834894
Title: Does Muscle Mass At Intensive Care Unit Admission Determine Mortality: the Memo Study
Acronym: MEMO
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: VBertoniMaluf (Unknown)
Responsible Party: Principal Investigator, Genton Graf Laurence, Prof., University Hospital, Geneva
Other Study IDs: 2022-01773
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Lean Body Mass
Keywords: Muscle mass; Skeletal muscle area; Third lumbar; Tomography; Intensive care unit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: exposure(s) of interest : intensive care unit — Low muscle mass is highly prevalent at hospital admission, and muscle mass generally decreases during hospital stay, especially in critically-ill patients. We would like to mesure muscle mas in critically ill patients and determine the association between outcomes.

SUMMARY:
This retrospective monocentric study aims to investigate whether a low muscle mass at ICU admission and its loss over the ICU stay predicts mortality, and in what proportion we can counteract it by nutritional support.

DETAILED DESCRIPTION:
The study hypothesis is that a low muscle mass at ICU admission, measured at the level of L3 on CT scans performed for clinical routine, and its change over the ICU stay predict the prognosis of the patient, especially the 30-day mortality, that it may at least be partly counteracted by nutritional support and that it is related with higher ICU and hospital costs.

The objectives of this retrospective study are to determine:

1. the link between baseline body composition at ICU admission and outcomes, such as 30-day, ICU and hospital mortality and LOS, and infections. If this is confirmed, we aim to evaluate the added values of body composition to ICU severity scores to predict 30-day mortality
2. the link between baseline body composition vs. other locations to predict outcomes
3. the impact of body composition changes on the afore-mentioned outcomes. If this is confirmed, we aim to evaluate the added value of changes in body composition to changes in ICU severity scores to predict 30-day mortality
4. the impact of nutritional support on body composition changes

ELIGIBILITY:
Inclusion Criteria:

* Associations of baseline body composition with clinical outcomes:

Adults ≥ 18 yrs, hospitalized in the ICU of the HUG between January 1st 2010 and December 31st 2022 and Abdominal, or thoraco-abdominal CT scan measured 48 hours before to 96 hours after ICU admission in the HUG

* Associations of body composition changes with clinical outcomes, nutritional support or medico-economic paratemers:

Identical as for the associations of baseline body composition with clinical outcomes and At least one additional CT performed during the hospital stay

Exclusion Criteria:

* Associations of baseline body composition with clinical outcomes:

CT scans of low quality or CT scans performed outside of the HUG or Presence of a documented refusal

* Associations of body composition changes with clinical outcomes, nutritional support or medico-economic paratemers:

Additionnally: oral nutrition, because we cannot assess the quantity and composition of oral intakes retrospectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ≥ 18 yrs, hospitalized in the ICU of the HUG between January 1st 2010 and December 31st 2022
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30-day mortality between January 1st 2010 and December 31st 2022.
  Association between skeletal muscle index (SMI) at the L3 vertebra level (psoas + abdominal wall muscles + paraspinal muscles), measured from 48 hours before to 96 hours after ICU admission, with 30-day mortality.

SECONDARY OUTCOMES:
Association of baseline body composition at ICU admission with other outcomes | 30-day
  Association of Skeletal muscle area (SMA), SMAH (Skeletal muscle area/height), SMD (Skeletal muscle density), IMAT (intermuscular and intramuscular adipose tissue), visceral and subcutaneous adipose tissue at the L3 vertebra level with 30-day mortality Determination of cut-off points of SMI, by sex, below which there is an increased risk of 30-day mortality Added value of body composition to ICU severity scores to predict 30-day mortality Association of baseline SMI, SMA, SMAH, SMD, intermuscular, visceral and subcutaneous adipose tissue at the L3 level, with ICU and hospital mortality and LOS, 30-day ICU readmission, duration of mechanical ventilation and infections
Association of baseline SMI at the L3 vertebra level vs. other locations to predict outcomes | Day 1 to day 30
  Associations of SMI at the L3 vertebra level with SMI at the other locations Associations of SMI at the other locations with ICU and hospital mortality and LOS, 30-day ICU readmission, duration of mechanical ventilation and infections Comparison of the associations between muscle mass measured at the different anatomical locations and mortality in order to determine the best prognostic location
Association of body composition changes with outcomes | Day 30
  Association of changes in SMI, SMA, SMAH, SMD, IMAT, visceral and subcutaneous adipose tissue with 30-day mortality, ICU and hospital mortality and LOS, 30-day ICU readmission, duration of mechanical ventilation and infections Added value of changes in body composition to changes in ICU severity scores to predict 30-day mortality
Association of body composition changes with nutritional support | Day 30
  Association of changes in energy coverage and changes in body composition Association of changes in protein coverage and changes in body composition
Association of muscle loss with medico-economical parameters | Day 30
  Association of baseline muscle mass and muscle loss in the ICU with ICU and hospital costs Association of muscle loss in the ICU with level of nursing workload

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Genton, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Laurence Genton, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
IPD Sharing Plan Description has not been decided.

REFERENCES:
- [Derived] Genton L, Bertoni Maluf VA, Herrmann FR, Prado CM, de Watteville A, Dupertuis YM, Collet TH, Platon A, Heidegger CP. Obesity is associated with lower 30-day mortality in critically ill patients: A retrospective study of over 5400 patients. Clin Nutr ESPEN. 2025 Oct;69:37-44. doi: 10.1016/j.clnesp.2025.06.046. Epub 2025 Jun 30. PMID 40602605